CLINICAL TRIAL: NCT02490306
Title: An Open Multicentre Trial on Suspected Stroke Patients Evaluating the Possibility to Use Microwave Technology to Differentiate Hemorrhage From Infarction in the Acute Phase
Brief Title: Evaluating Use of Microwave Technology to Differentiate Hemorrhagic Stroke From Infarction in the Acute Phase
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mikael Elam (Other)
Collaborators: Medfield Diagnostics (Industry); Chalmers University of Technology (Other)
Responsible Party: Sponsor-Investigator, Mikael Elam, Professor, MD, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VGR 01
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hemorrhagic stroke (Experimental): Patient group A is defined as patients that are diagnosed with hemorrhagic stroke.
  Interventions: Strokefinder MD100 measurement
  Interventions: Device: Strokefinder MD100 measurement
- Ischemic stroke (Experimental): Patient group B is defined as patients that are diagnosed with ischemic stroke.
  Interventions: Strokefinder MD100 measurement
  Interventions: Device: Strokefinder MD100 measurement
- Stroke mimics (Experimental): Patient group C is defined as patients with stroke mimics, i.e. with initially suspected stroke but not diagnosed with stroke.
  Interventions: Strokefinder MD100 measurement
  Interventions: Device: Strokefinder MD100 measurement

INTERVENTIONS:
Device: Strokefinder MD100 measurement — A microwave measurement will be performed with the patient lying in the hospital bed or another suitable surface. Follow-up microwave measurements will be performed after the acute phase.

SUMMARY:
This is a prospective, open, multicentre trial that will enrol patients with clinical signs of stroke in the acute phase admitted for CT scan. Follow-up microwave measurements will be performed after the acute phase. The study assesses the diagnostic capability and safety of Strokefinder MD100.

DETAILED DESCRIPTION:
This is a prospective, open, multicentre trial that will enrol patients with clinical signs of stroke in the acute phase admitted for CT scan. The investigator will assess and control the inclusion/exclusion criteria. If the patient is confirmed to be suitable for the trial, the patient is asked to give oral informed consent. If the answer is affirmative the microwave measurement will be performed. The procedure will take less than five minutes (the duration of the actual measurement procedure is 1.5 minutes) and will not interfere with the patient's standard of care during the hospital stay. Written informed consent is acquired by the investigator, as soon as possible after the acute phase of care is completed. Follow-up microwave measurements will be performed after the acute phase.

The measurement data will be evaluated for the presence of signal artifacts. The diagnostic ability of the device will be evaluated using a leave-one-out cross validation (LOOCV) method with the CT diagnosis as ground truth.

Safety will be evaluated throughout the trial, and a safety follow-up will be performed by the investigator 24 hours after the last microwave measurement. No further follow-up of patients is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patient should be ≥ 18 years of age
* Patient has clinical signs of stroke
* Patient/next of kin confirms orally that the patient wants to participate in the trial (during acute phase)
* Signed Informed Consent Form (after acute phase)

Exclusion Criteria:

* Pregnant or nursing woman
* Fertile woman where pregnancy cannot be excluded
* Patient diagnosed with a condition associated with risk of poor protocol compliance
* The diagnostic procedure is deemed to interfere with the standard of care
* Any other condition or symptoms preventing the patient from entering the study, according to the investigator´s judgment
* Any patient that according to the Declaration of Helsinki is deemed unsuitable for study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-07; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The diagnostic ability as measured by the area under receiver operating characteristic curve (AUC) of the device for patient group A vs. group B, using the leave-one-out cross validation (LOOCV) method | The diagnostic procedure will take less than 5 minutes

SECONDARY OUTCOMES:
The diagnostic ability as measured by the AUC of the device for patient group C vs. groups A + B, using the LOOCV method | The diagnostic procedure will take less than 5 minutes
Any adverse events occurring within 24 hours from the measurement procedure(s) | Within 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Elam, PhD, MD, Principal Investigator — Sahlgrenska University Hospital, Department of Clinical Neurophysiology
Locations (1):
- Sahlgrenska University Hospital, Stroke Unit, Gothenburg, Västra Götaland County, Sweden